CLINICAL TRIAL: NCT00799903
Title: LPL100601, A Clinical Outcomes Study of Darapladib Versus Placebo in Subjects With Chronic Coronary Heart Disease to Compare the Incidence of Major Adverse Cardiovascular Events (MACE)
Brief Title: The Stabilization of Atherosclerotic Plaque by Initiation of Darapladib Therapy Trial
Acronym: STABILITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100601
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-03

CONDITIONS: Atherosclerosis
Keywords: heart disease; Lp-PLA2 inhibitor; cardiovascular disease; coronary heart disease; CV risk; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Heart Diseases; Cardiovascular Diseases; Coronary Disease | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darapladib (Experimental): Single daily oral tablet
  Interventions: Drug: Darapladib
- Placebo (Placebo Comparator): Single daily oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darapladib — Lp-PLA2 inhibitor administered in addition to standard therapy
  Arms: Darapladib
Drug: Placebo — Placebo administered in addition to standard therapy
  Arms: Placebo

SUMMARY:
This study will test whether darapladib can safely lower the chances of having a cardiovascular event (such as a heart attack or stroke) in people with coronary heart disease.

DETAILED DESCRIPTION:
Subjects who qualify for the study will be randomized 1:1 to either darapladib or placebo administered in addition to standard therapy. Following the baseline visit, subjects will be expected to return for clinic visits at 1 month, 3 months, and every 6 months until the end of the study. Average time in the study for an individual subject is expected to be about 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years old. Women must be post-menopausal or using a highly effective method for avoidance of pregnancy.
* Current treatment with statin therapy unless the study doctor determines statins are not appropriate for the subject.
* Chronic coronary heart disease
* At least one of the following:
* At least 60 years old
* Diabetes requiring treatment with medication
* Low HDL cholesterol ("good cholesterol")
* Currently smoke cigarettes or stopped smoking within the past 3 months
* Diagnosed mild or moderate reduction in kidney function
* Cerebrovascular disease (carotid artery disease or ischemic stroke more than 3 months prior to study entry) OR peripheral arterial disease.

Exclusion Criteria:

* Planned coronary revascularization (such as stent placement or heart bypass) or any other major surgical procedure.
* Liver disease
* Severe reduction in kidney function OR removal of a kidney OR kidney transplant
* Severe heart failure
* Blood pressure higher than normal despite lifestyle changes and treatment with medications
* Any life-threatening disease expected to result in death within the next 2 years (other than heart disease)
* Severe asthma that is poorly controlled with medication
* Pregnant (Note: A pregnancy test will be performed on all non-sterile women prior to study entry)
* Previous severe allergic response to food, drink, insect stings, etc.
* Drug or alcohol abuse within the past 6 months OR mental/psychological impairment that may prevent the subject from complying with study procedures or understanding the goal and potential risks of participating in the study.
* Certain medications that may interfere with the study medication (these will be identified by the study doctor)
* Participation in a study of an investigational medication within the past 30 days
* Current participation in a study of an investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15828 (Actual)
Dates: Start 2008-12-01; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (525):
- United States (135):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Thousand Oaks, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jacksonville Beach, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Ponte Vedra Beach, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Franklin, Indiana
  - GSK Investigational Site, Greenfield, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Iberia, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Prince Frederick, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Natick, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Petoskey, Michigan
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Browns Mills, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Elyria, Ohio
  - GSK Investigational Site, Garfield Heights, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Sandusky, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Westlake, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Danville, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Jersey Shore, Pennsylvania
  - GSK Investigational Site, Lewistown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Philipsburg, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Port Matilda, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Scranton, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Wilkes-Barre, Pennsylvania
  - GSK Investigational Site, York, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Harker Heights, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Victoria, Texas
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Olympia, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Wausau, Wisconsin
- Argentina (16):
  - GSK Investigational Site, Adrogué, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Junín, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Ramos Mejía, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Australia (16):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Ballarat, Victoria
  - GSK Investigational Site, Caulfield South, Victoria
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Joondalup, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (11):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselaere
  - GSK Investigational Site, Yvoir
- Brazil (11):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Natal, Rio Grande do Norte
  - GSK Investigational Site, Pelotas, Rio Grande do Sul
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Bulgaria (6):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Veliko Tarnovo
- Canada (29):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Talcahuano, Región Del Biobio
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Haerbin
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan
- Czechia (15):
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Chrudim
  - GSK Investigational Site, Čáslav
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Kolín
  - GSK Investigational Site, Kroměříž
  - GSK Investigational Site, Milevsko
  - GSK Investigational Site, Písek
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Příbram
  - GSK Investigational Site, Slaný
  - GSK Investigational Site, Svitavy
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Ústí nad Orlicí
- Denmark (4):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Koebenhavn OE
  - GSK Investigational Site, Silkeborg
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (18):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Narbonne
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Roubaix
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
- Germany (35):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Mühldorf, Bavaria
  - GSK Investigational Site, Sulzbach-Rosenberg, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Bernau bei Berlin, Brandenburg
  - GSK Investigational Site, Frankfurt/M., Hesse
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Weyhe-Leeste, Lower Saxony
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Dorsten, North Rhine-Westphalia
  - GSK Investigational Site, Eschweiler, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Herford, North Rhine-Westphalia
  - GSK Investigational Site, Lienen-Kattenvenne, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (9):
  - GSK Investigational Site, Agia Varvara, Athens
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chalcis
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Magoula, Elefsina
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Voula / Athens
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin, New Territories
- Hungary (10):
  - GSK Investigational Site, Berettyóújfalu
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Esztergom
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Komárom
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Sátoraljaújhely
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szikszó
  - GSK Investigational Site, Szolnok
- India (11):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Mysore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Patiāla
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Saket,Delhi
  - GSK Investigational Site, Vadodara
  - GSK Investigational Site, Vijayawada
- Italy (12):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Carpi, Emilia-Romagna
  - GSK Investigational Site, Cona (Ferrara), Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Ascoli Piceno, The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Treviso, Veneto
- Japan (14):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Durango
  - GSK Investigational Site, México
  - GSK Investigational Site, México D.F,
- Netherlands (14):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Beverwijk
  - GSK Investigational Site, Doetinchem
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Goes
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tiel
- New Zealand (12):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Grafton, Auckland
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Nelson
  - GSK Investigational Site, Otahuhu, Auckland
  - GSK Investigational Site, Palmerston North
  - GSK Investigational Site, Takapuna, Auckland
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Timaru
  - GSK Investigational Site, Whangarei
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Moss
  - GSK Investigational Site, Oslo
- Pakistan (5):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Korangi / Karachi
  - GSK Investigational Site, Lahore
  - GSK Investigational Site, Multan
  - GSK Investigational Site, Rawalpindi Cantt
- Peru (3):
  - GSK Investigational Site, Jesus Maria, Lima region
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Philippines (4):
  - GSK Investigational Site, Ermita, Manila
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
- Poland (16):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Kowanówko
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Mielec
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Płońsk
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Tychy
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Włocławek
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Târgu Mureş
- Russia (9):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, S.-Petresburg
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Yekaterinburg
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Nitra
- South Africa (14):
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Kuils River
  - GSK Investigational Site, Moreletapark
  - GSK Investigational Site, Olivedale
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Parktown West
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Pinelands
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Soweto
  - GSK Investigational Site, Umhlanga
- South Korea (9):
  - GSK Investigational Site, Cheongju-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gangnam-gu, Seoul
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Jeonju-si, Jeollabuk-Do
  - GSK Investigational Site, Seo-gu Busan
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Uijeongbu-si Kyonggi-do
- Spain (15):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, San Juan (Alicante)
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, San Sebastián de Los Reyes/Madrid
  - GSK Investigational Site, Santa Coloma de Gramanet (Barcelona)
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valdemoro/Madrid
- Sweden (11):
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Västerås
  - GSK Investigational Site, Västervik
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Ukraine (7):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia
- United Kingdom (17):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Motherwell, Lanarkshire
  - GSK Investigational Site, Chelsea, London
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Chertsey, Surrey
  - GSK Investigational Site, Chichester, Sussex West
  - GSK Investigational Site, Barnet
  - GSK Investigational Site, Coatbridge
  - GSK Investigational Site, Cottingham
  - GSK Investigational Site, Cumbernauld
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Hertfordshire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Paisley

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jiang W, Huang G, Du J, Yang H, Zhou S, Dai D, Tang K, Fang L, Wang X, Deng X. White blood cell counts can predict 4-year cardiovascular disease risk in patients with stable coronary heart disease: a prospective cohort study. Front Cardiovasc Med. 2024 Sep 26;11:1358378. doi: 10.3389/fcvm.2024.1358378. eCollection 2024. PMID 39390990
- [Derived] Sjolin K, Aulin J, Wallentin L, Eriksson N, Held C, Kultima K, Oldgren J, Burman J. Serum Neurofilament Light Chain in Patients With Atrial Fibrillation. J Am Heart Assoc. 2022 Jul 19;11(14):e025910. doi: 10.1161/JAHA.122.025910. Epub 2022 Jul 15. PMID 35861814
- [Derived] Held C, Hadziosmanovic N, Aylward PE, Hagstrom E, Hochman JS, Stewart RAH, White HD, Wallentin L. Body Mass Index and Association With Cardiovascular Outcomes in Patients With Stable Coronary Heart Disease - A STABILITY Substudy. J Am Heart Assoc. 2022 Feb;11(3):e023667. doi: 10.1161/JAHA.121.023667. Epub 2022 Jan 21. PMID 35060389
- [Derived] Siddiqui MK, Smith G, St Jean P, Dawed AY, Bell S, Soto-Pedre E, Kennedy G, Carr F, Wallentin L, White H, Macphee CH, Waterworth D, Palmer CNA. Diabetes status modifies the long-term effect of lipoprotein-associated phospholipase A2 on major coronary events. Diabetologia. 2022 Jan;65(1):101-112. doi: 10.1007/s00125-021-05574-5. Epub 2021 Sep 25. PMID 34562103
- [Derived] Wallentin L, Eriksson N, Olszowka M, Grammer TB, Hagstrom E, Held C, Kleber ME, Koenig W, Marz W, Stewart RAH, White HD, Aberg M, Siegbahn A. Plasma proteins associated with cardiovascular death in patients with chronic coronary heart disease: A retrospective study. PLoS Med. 2021 Jan 13;18(1):e1003513. doi: 10.1371/journal.pmed.1003513. eCollection 2021 Jan. PMID 33439866
- [Derived] White HD, Stewart RAH, Dalby AJ, Stebbins A, Cannon CP, Budaj A, Linhart A, Pais P, Diaz R, Steg PG, Krug-Gourley S, Granger CB, Hochman JS, Koenig W, Harrington RA, Held C, Wallentin L; STABILITY Investigators. In patients with stable coronary heart disease, low-density lipoprotein-cholesterol levels < 70 mg/dL and glycosylated hemoglobin A1c < 7% are associated with lower major cardiovascular events. Am Heart J. 2020 Jul;225:97-107. doi: 10.1016/j.ahj.2020.04.004. Epub 2020 Apr 18. PMID 32480059
- [Derived] Hilvo M, Wallentin L, Ghukasyan Lakic T, Held C, Kauhanen D, Jylha A, Lindback J, Siegbahn A, Granger CB, Koenig W, Stewart RAH, White H, Laaksonen R; STABILITY Investigators. Prediction of Residual Risk by Ceramide-Phospholipid Score in Patients With Stable Coronary Heart Disease on Optimal Medical Therapy. J Am Heart Assoc. 2020 May 18;9(10):e015258. doi: 10.1161/JAHA.119.015258. Epub 2020 May 7. PMID 32375553
- [Derived] Stewart RAH, Held C, Krug-Gourley S, Waterworth D, Stebbins A, Chiswell K, Hagstrom E, Armstrong PW, Wallentin L, White H. Cardiovascular and Lifestyle Risk Factors and Cognitive Function in Patients With Stable Coronary Heart Disease. J Am Heart Assoc. 2019 Apr 2;8(7):e010641. doi: 10.1161/JAHA.118.010641. PMID 30897999
- [Derived] Held C, White HD, Stewart RAH, Budaj A, Cannon CP, Hochman JS, Koenig W, Siegbahn A, Steg PG, Soffer J, Weaver WD, Ostlund O, Wallentin L; STABILITY Investigators. Inflammatory Biomarkers Interleukin-6 and C-Reactive Protein and Outcomes in Stable Coronary Heart Disease: Experiences From the STABILITY (Stabilization of Atherosclerotic Plaque by Initiation of Darapladib Therapy) Trial. J Am Heart Assoc. 2017 Oct 24;6(10):e005077. doi: 10.1161/JAHA.116.005077. PMID 29066452
- [Derived] Hagstrom E, Norlund F, Stebbins A, Armstrong PW, Chiswell K, Granger CB, Lopez-Sendon J, Pella D, Soffer J, Sy R, Wallentin L, White HD, Stewart RAH, Held C. Psychosocial stress and major cardiovascular events in patients with stable coronary heart disease. J Intern Med. 2018 Jan;283(1):83-92. doi: 10.1111/joim.12692. Epub 2017 Oct 23. PMID 28960596
- [Derived] Guimaraes PO, Granger CB, Stebbins A, Chiswell K, Held C, Hochman JS, Krug-Gourley S, Lonn E, Lopes RD, Stewart RAH, Vinereanu D, Wallentin L, White HD, Hagstrom E, Danchin N. Sex Differences in Clinical Characteristics, Psychosocial Factors, and Outcomes Among Patients With Stable Coronary Heart Disease: Insights from the STABILITY (Stabilization of Atherosclerotic Plaque by Initiation of Darapladib Therapy) Trial. J Am Heart Assoc. 2017 Sep 14;6(9):e006695. doi: 10.1161/JAHA.117.006695. PMID 28912210
- [Derived] Stewart RAH, Hagstrom E, Held C, Wang TKM, Armstrong PW, Aylward PE, Cannon CP, Koenig W, Lopez-Sendon JL, Mohler ER 3rd, Hadziosmanovic N, Krug-Gourley S, Ramos Corrales MA, Siddique S, Steg PG, White HD, Wallentin L; STABILITY Investigators. Self-Reported Health and Outcomes in Patients With Stable Coronary Heart Disease. J Am Heart Assoc. 2017 Aug 22;6(8):e006096. doi: 10.1161/JAHA.117.006096. PMID 28862971
- [Derived] Lindholm D, Lindback J, Armstrong PW, Budaj A, Cannon CP, Granger CB, Hagstrom E, Held C, Koenig W, Ostlund O, Stewart RAH, Soffer J, White HD, de Winter RJ, Steg PG, Siegbahn A, Kleber ME, Dressel A, Grammer TB, Marz W, Wallentin L. Biomarker-Based Risk Model to Predict Cardiovascular Mortality in Patients With Stable Coronary Disease. J Am Coll Cardiol. 2017 Aug 15;70(7):813-826. doi: 10.1016/j.jacc.2017.06.030. PMID 28797349
- [Derived] Vedin O, Hagstrom E, Ostlund O, Avezum A, Budaj A, Flather MD, Harrington RA, Koenig W, Soffer J, Siegbahn A, Steg PG, Stewart RAH, Wallentin L, White HD, Held C; STABILITY Investigators. Associations between tooth loss and prognostic biomarkers and the risk for cardiovascular events in patients with stable coronary heart disease. Int J Cardiol. 2017 Oct 15;245:271-276. doi: 10.1016/j.ijcard.2017.07.036. Epub 2017 Jul 17. PMID 28735759
- [Derived] Hagstrom E, Held C, Stewart RA, Aylward PE, Budaj A, Cannon CP, Koenig W, Krug-Gourley S, Mohler ER 3rd, Steg PG, Tarka E, Ostlund O, White HD, Siegbahn A, Wallentin L; STABILITY Investigators. Growth Differentiation Factor 15 Predicts All-Cause Morbidity and Mortality in Stable Coronary Heart Disease. Clin Chem. 2017 Jan;63(1):325-333. doi: 10.1373/clinchem.2016.260570. Epub 2016 Nov 3. PMID 27811204
- [Derived] Wallentin L, Held C, Armstrong PW, Cannon CP, Davies RY, Granger CB, Hagstrom E, Harrington RA, Hochman JS, Koenig W, Krug-Gourley S, Mohler ER 3rd, Siegbahn A, Tarka E, Steg PG, Stewart RA, Weiss R, Ostlund O, White HD; STABILITY Investigators. Lipoprotein-Associated Phospholipase A2 Activity Is a Marker of Risk But Not a Useful Target for Treatment in Patients With Stable Coronary Heart Disease. J Am Heart Assoc. 2016 Jun 21;5(6):e003407. doi: 10.1161/JAHA.116.003407. PMID 27329448
- [Derived] Hijazi Z, Lindback J, Alexander JH, Hanna M, Held C, Hylek EM, Lopes RD, Oldgren J, Siegbahn A, Stewart RA, White HD, Granger CB, Wallentin L; ARISTOTLE and STABILITY Investigators. The ABC (age, biomarkers, clinical history) stroke risk score: a biomarker-based risk score for predicting stroke in atrial fibrillation. Eur Heart J. 2016 May 21;37(20):1582-90. doi: 10.1093/eurheartj/ehw054. Epub 2016 Feb 25. PMID 26920728
- [Derived] Vedin O, Hagstrom E, Budaj A, Denchev S, Harrington RA, Koenig W, Soffer J, Sritara P, Stebbins A, Stewart RH, Swart HP, Viigimaa M, Vinereanu D, Wallentin L, White HD, Held C; STABILITY Investigators. Tooth loss is independently associated with poor outcomes in stable coronary heart disease. Eur J Prev Cardiol. 2016 May;23(8):839-46. doi: 10.1177/2047487315621978. Epub 2015 Dec 16. PMID 26672609
- [Derived] Vedin O, Hagstrom E, Gallup D, Neely ML, Stewart R, Koenig W, Budaj A, Sritara P, Wallentin L, White HD, Held C. Periodontal disease in patients with chronic coronary heart disease: Prevalence and association with cardiovascular risk factors. Eur J Prev Cardiol. 2015 Jun;22(6):771-8. doi: 10.1177/2047487314530660. Epub 2014 Apr 10. PMID 24721691
- [Derived] STABILITY Investigators; White HD, Held C, Stewart R, Tarka E, Brown R, Davies RY, Budaj A, Harrington RA, Steg PG, Ardissino D, Armstrong PW, Avezum A, Aylward PE, Bryce A, Chen H, Chen MF, Corbalan R, Dalby AJ, Danchin N, De Winter RJ, Denchev S, Diaz R, Elisaf M, Flather MD, Goudev AR, Granger CB, Grinfeld L, Hochman JS, Husted S, Kim HS, Koenig W, Linhart A, Lonn E, Lopez-Sendon J, Manolis AJ, Mohler ER 3rd, Nicolau JC, Pais P, Parkhomenko A, Pedersen TR, Pella D, Ramos-Corrales MA, Ruda M, Sereg M, Siddique S, Sinnaeve P, Smith P, Sritara P, Swart HP, Sy RG, Teramoto T, Tse HF, Watson D, Weaver WD, Weiss R, Viigimaa M, Vinereanu D, Zhu J, Cannon CP, Wallentin L. Darapladib for preventing ischemic events in stable coronary heart disease. N Engl J Med. 2014 May 1;370(18):1702-11. doi: 10.1056/NEJMoa1315878. Epub 2014 Mar 30. PMID 24678955
- [Derived] Vedin O, Hagstrom E, Stewart R, Brown R, Krug-Gourley S, Davies R, Wallentin L, White H, Held C. Secondary prevention and risk factor target achievement in a global, high-risk population with established coronary heart disease: baseline results from the STABILITY study. Eur J Prev Cardiol. 2013 Aug;20(4):678-85. doi: 10.1177/2047487312444995. Epub 2012 Apr 10. PMID 22496275
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a Screening Phase of up to 8 weeks duration, a Treatment Phase, an End-of-Treatment (EOT) visit, and a Follow-up visit scheduled for 35 +/- 7 days after last study drug intake. The median treatment duration was anticipated to be 2.75 years.
Pre-assignment Details: During the Screening Phase of the study, participants presenting with chronic Coronary Heart Disease (CHD) were randomized within 8 weeks. In addition to chronic CHD, participants were required to have at least one additional predictor of cardiovascular risk specified in the protocol.
Groups:
- Placebo: Participants were randomized to receive matching placebo once daily.
- Darapladib: Participants were randomized to receive darapladib 160 milligram (mg) enteric-coated tablets once daily.
Period: Overall Study
Arm/Group | Placebo | Darapladib
Started | 7904 | 7924
Completed | 7631 | 7646
Not Completed | 273 | 278
Not completed — Investigator Site Closed | 25 | 23
Not completed — Withdrawal by Subject | 179 | 175
Not completed — Lost to Follow-up | 69 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Darapladib | Total
Number analyzed (Participants) | 7904 | 7924 | 15828
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.39) | 64.5 (9.31) | 64.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1506 | 1461 | 2967
  Male | 6398 | 6463 | 12861
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 108 | 106 | 214
  Asian | 1366 | 1351 | 2717
  Native Hawaiian or Other Pacific Islander | 11 | 4 | 15
  Black or African American | 191 | 175 | 366
  White | 6177 | 6233 | 12410
  More than one race | 51 | 55 | 106
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Any Component of the Composite of Major Adverse Cardiovascular Events (Cardiovascular [CV] Death, Non-fatal Myocardial Infarction [MI] or Non-fatal Stroke) During the Time Period for Follow-up of CV Events
Description: CV death=death due to a CV cause, which included but was not limited to deaths resulting from stroke, arrhythmia, sudden death (witnessed/unwitnessed), MI, heart failure, pulmonary embolism, peripheral arterial disease, or complications of a CV procedure. Deaths not clearly attributable to non-CV causes are considered to be CV deaths. Acute MI=evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Stroke=presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: From randomization until the End-of-Treatment visit or the last date on which endpoints were able to be assessed (up to 4.25 years/average of 3.51 years)
Population: All-randomized Intent-to-treat (ITT) population comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 819 | 769
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.199, Regression, Cox — Hazard ratio and p-value are estimated using a Cox proportional hazard regression model with treatment as the only covariate. A hazard ratio < 1 indicates a lower risk with this treatment compared to Placebo; Hazard Ratio (HR) = 0.94, 95.1% CI 2-sided [0.85 to 1.03]

2. Secondary Outcome: Number of Participants With First Occurrence of Any Event in the Composite of Major Coronary Events (Coronary Heart Disease [CHD] Death, Non-fatal MI, or Urgent Coronary Revascularization [CR] for MI) During the Time Period for Follow-up (FU) of CV Events
Description: CHD death=occurrence of a fatal MI, death caused by documented cardiac arrest, death resulting from heart failure in a participant with known CHD, death from other forms of acute/chronic CHD, unwitnessed death of unknown origin, or sudden death. Acute MI=evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g.,silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Urgent CR for MI=ischemic discomfort at rest that prompted CR (percutaneous coronary intervention [PCI: any attempt at CR even if not successful] or coronary artery bypass graft) during the same hospitalization or resulted in hospital transfer for the purpose of CR.
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 814 | 737
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.045, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.82 to 1.00]

3. Secondary Outcome: Number of Participants With First Occurrence of Any Event in the Composite of Total Coronary Events (CHD Death, Non-fatal MI, Hospitalization for Unstable Angina, or Any Coronary Revascularization Procedure) During Time Period for FU of CV Events
Description: CHD death, acute MI, and prior MI are defined in the previous secondary endpoint (major coronary events). Hospitalization for unstable angina=one of the following, but not fulfilling the criteria for MI: ischemic discomfort at rest associated with electrocardiogram (ECG) changes leading to hospitalization; ischemic discomfort at rest regardless of ECG changes leading to hospitalization and revascularization during the same admission; ischemic discomfort at rest in hospital associated with ECG changes; ischemic discomfort at rest in hospital without ECG changes resulting in revascularization during the same admission. NOTE: The event was not considered to be unstable angina if, after invasive/non-invasive testing or other diagnostic testing, the discomfort is found not to be caused by myocardial ischemia.
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 1269 | 1159
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.019, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.84 to 0.98]

4. Secondary Outcome: Number of Participants With CV Death During the Time Period for Follow-up of CV Events
Description: CV death is defined as a death due to a CV cause, which included but was not limited to deaths resulting from stroke, arrhythmia, sudden death (witnessed/unwitnessed), MI, heart failure, pulmonary embolism, peripheral arterial disease, or complications of a CV procedure. Deaths not clearly attributable to non-CV causes are considered to be CV deaths.
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 373 | 359
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.594, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.83 to 1.11]

5. Secondary Outcome: Number of Participants With First Occurrence of MI (Fatal/Non-fatal) During the Time Period for Follow-up of CV Events
Description: Acute MI is defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI.
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 405 | 361
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.108, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.03]

6. Secondary Outcome: Number of Participants With First Occurrence of Stroke (Fatal/Non-fatal) During the Time Period for Follow-up of CV Events
Description: Stroke is defined as the presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 152 | 154
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.920, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.81 to 1.27]

7. Secondary Outcome: Number of Participants With First Occurrence of Any Component of the Composite of All-cause Mortality, Non-fatal MI, or Non-fatal Stroke During the Time Period for Follow-up of CV Events
Description: Acute MI is defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Stroke=presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: as for outcome 1
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 962 | 926
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.397, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.88 to 1.05]

8. Secondary Outcome: Number of Participants With All-cause Mortality During the Time Period for Vital Status
Description: The number of participants with all-cause mortality was assessed.
Time Frame: From randomization until death or study completion (up to 4.49 years/average of 3.65 years)
Population: All Randomized (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib
Number analyzed (Participants) | 7904 | 7924
Participants | 577 | 582
Statistical Analysis 1: Comparison: Placebo vs Darapladib; Test type: Superiority; p = 0.870, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.90 to 1.13]

ADVERSE EVENTS:
Time Frame: Start=Randomization; Stop=Longer of 35 days after last dose of IP or follow-up (FU) visit. "SAEs assessed as related to IP, study participation, or a GSK concomitant medication" and cancer/GI polyps/neoplasms were recorded up to/including any FU contact.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of investigational product. Post-randomization AEs have an onset date that is on or after the randomization date.
Arm/Group | Placebo | Darapladib
All-Cause Mortality (participants affected / at risk) | 577/7904 | 582/7924
Serious Adverse Events (participants affected / at risk) | 3448/7890 | 3369/7912
Other Adverse Events (participants affected / at risk) | 4885/7890 | 5171/7912
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7890) | Darapladib (N=7912)
Angina unstable (Cardiac disorders) | 489 | 472
Acute myocardial infarction (Cardiac disorders) | 359 | 303
Angina pectoris (Cardiac disorders) | 271 | 248
Coronary artery disease (Cardiac disorders) | 177 | 168
Cardiac failure (Cardiac disorders) | 178 | 155
Cardiac failure congestive (Cardiac disorders) | 135 | 125
Atrial fibrillation (Cardiac disorders) | 135 | 123
Coronary artery stenosis (Cardiac disorders) | 59 | 56
Myocardial infarction (Cardiac disorders) | 54 | 56
Myocardial ischaemia (Cardiac disorders) | 41 | 47
Ventricular tachycardia (Cardiac disorders) | 42 | 37
Atrial flutter (Cardiac disorders) | 27 | 27
Cardiac arrest (Cardiac disorders) | 26 | 28
Bradycardia (Cardiac disorders) | 19 | 24
Ventricular fibrillation (Cardiac disorders) | 19 | 22
Sick sinus syndrome (Cardiac disorders) | 24 | 15
Cardiac failure chronic (Cardiac disorders) | 19 | 17
Coronary artery occlusion (Cardiac disorders) | 17 | 19
Acute coronary syndrome (Cardiac disorders) | 17 | 17
Cardio-respiratory arrest (Cardiac disorders) | 15 | 15
Cardiogenic shock (Cardiac disorders) | 11 | 16
Cardiac failure acute (Cardiac disorders) | 16 | 10
Ischaemic cardiomyopathy (Cardiac disorders) | 14 | 11
Supraventricular tachycardia (Cardiac disorders) | 8 | 14
Left ventricular dysfunction (Cardiac disorders) | 8 | 13
Arteriosclerosis coronary artery (Cardiac disorders) | 15 | 5
Mitral valve incompetence (Cardiac disorders) | 9 | 10
Left ventricular failure (Cardiac disorders) | 6 | 12
Aortic valve stenosis (Cardiac disorders) | 10 | 7
Atrioventricular block complete (Cardiac disorders) | 12 | 5
Ventricular extrasystoles (Cardiac disorders) | 9 | 8
Arrhythmia (Cardiac disorders) | 8 | 7
Atrioventricular block second degree (Cardiac disorders) | 7 | 8
Atrioventricular block (Cardiac disorders) | 9 | 5
Palpitations (Cardiac disorders) | 9 | 5
Cardiac discomfort (Cardiac disorders) | 6 | 5
Pericardial effusion (Cardiac disorders) | 6 | 5
Cardiovascular disorder (Cardiac disorders) | 6 | 4
Cardiopulmonary failure (Cardiac disorders) | 2 | 6
Cardiomyopathy (Cardiac disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 4 | 3
Atrial tachycardia (Cardiac disorders) | 1 | 5
Arrhythmia supraventricular (Cardiac disorders) | 4 | 1
Cardiac disorder (Cardiac disorders) | 3 | 2
Cardiovascular insufficiency (Cardiac disorders) | 4 | 1
Congestive cardiomyopathy (Cardiac disorders) | 4 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 4
Ventricular arrhythmia (Cardiac disorders) | 1 | 4
Bundle branch block left (Cardiac disorders) | 2 | 2
Cardiac asthma (Cardiac disorders) | 1 | 3
Right ventricular failure (Cardiac disorders) | 3 | 1
Acute left ventricular failure (Cardiac disorders) | 3 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 2
Arteriospasm coronary (Cardiac disorders) | 2 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 2
Cardiac tamponade (Cardiac disorders) | 2 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 2
Myocardial fibrosis (Cardiac disorders) | 2 | 1
Bradyarrhythmia (Cardiac disorders) | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Postinfarction angina (Cardiac disorders) | 2 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 2 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 2
Sinus arrest (Cardiac disorders) | 1 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 2
Stress cardiomyopathy (Cardiac disorders) | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 2
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve disease mixed (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Atrioventricular dissociation (Cardiac disorders) | 0 | 1
Bifascicular block (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiovascular deconditioning (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0
Chronotropic incompetence (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular dyssynchrony (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 160 | 139
Cellulitis (Infections and infestations) | 46 | 38
Urinary tract infection (Infections and infestations) | 36 | 43
Gastroenteritis (Infections and infestations) | 29 | 31
Sepsis (Infections and infestations) | 23 | 35
Bronchitis (Infections and infestations) | 18 | 24
Appendicitis (Infections and infestations) | 19 | 15
Septic shock (Infections and infestations) | 25 | 9
Urosepsis (Infections and infestations) | 15 | 14
Diverticulitis (Infections and infestations) | 11 | 15
Lobar pneumonia (Infections and infestations) | 17 | 9
Erysipelas (Infections and infestations) | 14 | 8
Bronchopneumonia (Infections and infestations) | 7 | 12
Localised infection (Infections and infestations) | 9 | 9
Lower respiratory tract infection (Infections and infestations) | 10 | 8
Pyelonephritis (Infections and infestations) | 6 | 12
Osteomyelitis (Infections and infestations) | 7 | 10
Respiratory tract infection (Infections and infestations) | 7 | 8
Device related infection (Infections and infestations) | 8 | 6
Influenza (Infections and infestations) | 7 | 7
Lung infection (Infections and infestations) | 8 | 5
Staphylococcal infection (Infections and infestations) | 6 | 6
Gastroenteritis viral (Infections and infestations) | 5 | 5
Herpes zoster (Infections and infestations) | 5 | 5
Peritonitis (Infections and infestations) | 7 | 3
Wound infection (Infections and infestations) | 6 | 3
Infection (Infections and infestations) | 4 | 4
Postoperative wound infection (Infections and infestations) | 3 | 5
Gangrene (Infections and infestations) | 4 | 3
Post procedural infection (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Appendicitis perforated (Infections and infestations) | 3 | 3
Bacteraemia (Infections and infestations) | 1 | 5
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 3
Viral infection (Infections and infestations) | 2 | 4
Abscess (Infections and infestations) | 5 | 0
Arthritis infective (Infections and infestations) | 2 | 3
Cholecystitis infective (Infections and infestations) | 1 | 4
Clostridium difficile infection (Infections and infestations) | 3 | 2
Pulmonary tuberculosis (Infections and infestations) | 3 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 4
Anal abscess (Infections and infestations) | 1 | 3
Arthritis bacterial (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 2 | 2
Diabetic gangrene (Infections and infestations) | 2 | 2
Endocarditis (Infections and infestations) | 0 | 4
Enterocolitis infectious (Infections and infestations) | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 3 | 1
Escherichia sepsis (Infections and infestations) | 0 | 4
Orchitis (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 4
Postoperative abscess (Infections and infestations) | 0 | 4
Skin infection (Infections and infestations) | 2 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 3
Abscess limb (Infections and infestations) | 2 | 1
Dengue fever (Infections and infestations) | 1 | 2
Diabetic foot infection (Infections and infestations) | 2 | 1
Enterococcal sepsis (Infections and infestations) | 2 | 1
H1N1 influenza (Infections and infestations) | 2 | 1
Haematoma infection (Infections and infestations) | 2 | 1
Intervertebral discitis (Infections and infestations) | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 2
Salmonellosis (Infections and infestations) | 1 | 2
Sepsis syndrome (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Streptococcal bacteraemia (Infections and infestations) | 1 | 2
Acute hepatitis B (Infections and infestations) | 1 | 1
Arteriosclerotic gangrene (Infections and infestations) | 1 | 1
Bacterial pyelonephritis (Infections and infestations) | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 1
Chronic sinusitis (Infections and infestations) | 2 | 0
Device related sepsis (Infections and infestations) | 1 | 1
Dysentery (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Extradural abscess (Infections and infestations) | 1 | 1
Gastritis viral (Infections and infestations) | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Giardiasis (Infections and infestations) | 2 | 0
Hepatitis B (Infections and infestations) | 2 | 0
Implant site infection (Infections and infestations) | 2 | 0
Infected skin ulcer (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 1 | 1
Lyme disease (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 2
Peritonsillar abscess (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia streptococcal (Infections and infestations) | 2 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 2 | 0
Retroperitoneal abscess (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 1 | 1
Streptococcal infection (Infections and infestations) | 2 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Acute pulmonary histoplasmosis (Infections and infestations) | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 1 | 0
Borrelia infection (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cholangitis suppurative (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Echinococciasis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Endocarditis enterococcal (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Genital infection fungal (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
HIV infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Infective myositis (Infections and infestations) | 0 | 1
Intertrigo candida (Infections and infestations) | 0 | 1
Keratitis herpetic (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Leptospirosis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0
Mycotoxicosis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Peritonsillitis (Infections and infestations) | 1 | 0
Plasmodium vivax infection (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyopneumothorax (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Retroperitoneal infection (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0
Scrub typhus (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinobronchitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subacute endocarditis (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 1 | 0
Suspected transmission of an infectious agent via product (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Tongue abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Tracheobronchitis viral (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Vaginal abscess (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral tracheitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 97 | 94
Transient ischaemic attack (Nervous system disorders) | 87 | 67
Syncope (Nervous system disorders) | 79 | 72
Carotid artery stenosis (Nervous system disorders) | 47 | 48
Cerebrovascular accident (Nervous system disorders) | 28 | 33
Dizziness (Nervous system disorders) | 18 | 18
Haemorrhagic stroke (Nervous system disorders) | 19 | 15
Ischaemic cerebral infarction (Nervous system disorders) | 20 | 13
Presyncope (Nervous system disorders) | 16 | 16
Cerebral infarction (Nervous system disorders) | 7 | 15
Convulsion (Nervous system disorders) | 8 | 5
Epilepsy (Nervous system disorders) | 5 | 7
Headache (Nervous system disorders) | 7 | 5
Sciatica (Nervous system disorders) | 6 | 6
Subarachnoid haemorrhage (Nervous system disorders) | 7 | 3
Brain stem infarction (Nervous system disorders) | 4 | 5
Embolic stroke (Nervous system disorders) | 4 | 5
Loss of consciousness (Nervous system disorders) | 4 | 5
Carotid artery occlusion (Nervous system disorders) | 7 | 1
Cervicobrachial syndrome (Nervous system disorders) | 4 | 4
Dementia (Nervous system disorders) | 4 | 4
Diabetic neuropathy (Nervous system disorders) | 4 | 4
Lacunar infarction (Nervous system disorders) | 6 | 2
Cerebral haemorrhage (Nervous system disorders) | 2 | 5
Carpal tunnel syndrome (Nervous system disorders) | 4 | 2
Haemorrhage intracranial (Nervous system disorders) | 3 | 3
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 2
Aphasia (Nervous system disorders) | 1 | 4
Carotid artery disease (Nervous system disorders) | 4 | 1
Embolic cerebral infarction (Nervous system disorders) | 3 | 2
Hemiparesis (Nervous system disorders) | 4 | 1
Tremor (Nervous system disorders) | 0 | 5
Ataxia (Nervous system disorders) | 3 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 3
Encephalopathy (Nervous system disorders) | 2 | 2
Metabolic encephalopathy (Nervous system disorders) | 1 | 3
Neuralgia (Nervous system disorders) | 2 | 2
VIIth nerve paralysis (Nervous system disorders) | 3 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 3
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Cognitive disorder (Nervous system disorders) | 1 | 2
Dysarthria (Nervous system disorders) | 2 | 1
Hypoglycaemic coma (Nervous system disorders) | 2 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 1 | 2
Polyneuropathy (Nervous system disorders) | 2 | 1
Thalamic infarction (Nervous system disorders) | 1 | 2
Vascular dementia (Nervous system disorders) | 2 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 2
Brain oedema (Nervous system disorders) | 1 | 1
Brain stem haemorrhage (Nervous system disorders) | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 2 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Intracranial aneurysm (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 1 | 1
Mononeuritis (Nervous system disorders) | 1 | 1
Nerve compression (Nervous system disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 1 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1
Paraplegia (Nervous system disorders) | 0 | 2
Post herpetic neuralgia (Nervous system disorders) | 1 | 1
Pseudoradicular syndrome (Nervous system disorders) | 0 | 2
Radiculopathy (Nervous system disorders) | 2 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 2 | 0
Senile dementia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0
Spondylitic myelopathy (Nervous system disorders) | 2 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 2 | 0
Transient global amnesia (Nervous system disorders) | 2 | 0
Vertebral artery stenosis (Nervous system disorders) | 1 | 1
Alcoholic seizure (Nervous system disorders) | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Brain midline shift (Nervous system disorders) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 1 | 0
Cerebral circulatory failure (Nervous system disorders) | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Critical illness polyneuropathy (Nervous system disorders) | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Diabetic mononeuropathy (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness exertional (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Dyslalia (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Encephalomalacia (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Hemianopia (Nervous system disorders) | 0 | 1
Hemiplegic migraine (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic neuropathy (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Meningoradiculitis (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Neuritis cranial (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Peripheral nerve paresis (Nervous system disorders) | 1 | 0
Polyneuropathy chronic (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Retrograde amnesia (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Simple partial seizures (Nervous system disorders) | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Spinal cord disorder (Nervous system disorders) | 1 | 0
Spinal haematoma (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Vascular parkinsonism (Nervous system disorders) | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
White matter lesion (Nervous system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 196 | 191
Death (General disorders) | 73 | 56
Sudden death (General disorders) | 56 | 57
Sudden cardiac death (General disorders) | 22 | 24
Chest pain (General disorders) | 18 | 11
Asthenia (General disorders) | 15 | 11
Pyrexia (General disorders) | 12 | 12
Device occlusion (General disorders) | 11 | 12
Fatigue (General disorders) | 9 | 8
Chest discomfort (General disorders) | 7 | 9
Oedema peripheral (General disorders) | 6 | 8
Multi-organ failure (General disorders) | 6 | 6
Device malfunction (General disorders) | 5 | 4
Hernia (General disorders) | 5 | 3
Malaise (General disorders) | 2 | 3
Medical device complication (General disorders) | 4 | 1
Device dislocation (General disorders) | 1 | 3
Adverse drug reaction (General disorders) | 2 | 1
Gait disturbance (General disorders) | 0 | 3
Thrombosis in device (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 2 | 0
Ill-defined disorder (General disorders) | 1 | 1
Medical device pain (General disorders) | 2 | 0
Pain (General disorders) | 1 | 1
Spinal pain (General disorders) | 1 | 1
Ulcer haemorrhage (General disorders) | 2 | 0
Axillary pain (General disorders) | 1 | 0
Cardiac complication associated with device (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Device battery issue (General disorders) | 1 | 0
Device lead damage (General disorders) | 0 | 1
Device lead issue (General disorders) | 1 | 0
Device power source issue (General disorders) | 1 | 0
Drowning (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fat necrosis (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site thrombosis (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Ischaemic ulcer (General disorders) | 1 | 0
Lipogranuloma (General disorders) | 1 | 0
Medical device site reaction (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 1 | 0
Nodule (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Stent embolisation (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vestibulitis (General disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 48 | 31
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 26 | 30
Diarrhoea (Gastrointestinal disorders) | 21 | 23
Abdominal pain (Gastrointestinal disorders) | 25 | 12
Large intestine polyp (Gastrointestinal disorders) | 16 | 21
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 | 14
Gastritis (Gastrointestinal disorders) | 18 | 12
Pancreatitis (Gastrointestinal disorders) | 15 | 15
Gastric ulcer (Gastrointestinal disorders) | 7 | 17
Nausea (Gastrointestinal disorders) | 12 | 11
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 13
Small intestinal obstruction (Gastrointestinal disorders) | 9 | 11
Colitis (Gastrointestinal disorders) | 12 | 7
Pancreatitis acute (Gastrointestinal disorders) | 12 | 7
Vomiting (Gastrointestinal disorders) | 12 | 7
Abdominal pain upper (Gastrointestinal disorders) | 7 | 11
Constipation (Gastrointestinal disorders) | 5 | 11
Intestinal obstruction (Gastrointestinal disorders) | 7 | 9
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 4
Ileus (Gastrointestinal disorders) | 7 | 6
Umbilical hernia (Gastrointestinal disorders) | 7 | 6
Diverticulum intestinal (Gastrointestinal disorders) | 5 | 7
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 7 | 5
Abdominal hernia (Gastrointestinal disorders) | 5 | 6
Colitis ischaemic (Gastrointestinal disorders) | 5 | 6
Duodenal ulcer (Gastrointestinal disorders) | 6 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6 | 5
Haemorrhoids (Gastrointestinal disorders) | 8 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 3 | 6
Gastritis erosive (Gastrointestinal disorders) | 7 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 5 | 4
Ascites (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 4 | 4
Melaena (Gastrointestinal disorders) | 3 | 5
Diverticulum (Gastrointestinal disorders) | 3 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 4 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 4 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 4
Gastritis haemorrhagic (Gastrointestinal disorders) | 3 | 2
Anal fistula (Gastrointestinal disorders) | 3 | 1
Enterovesical fistula (Gastrointestinal disorders) | 2 | 2
Haematemesis (Gastrointestinal disorders) | 2 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 4 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 3
Peptic ulcer (Gastrointestinal disorders) | 1 | 3
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2
Gastric polyps (Gastrointestinal disorders) | 2 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Large intestine perforation (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal strangulated hernia (Gastrointestinal disorders) | 2 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 1
Gastritis atrophic (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal angidysplasia (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 2
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 2 | 0
Stomach mass (Gastrointestinal disorders) | 1 | 1
Volvulus (Gastrointestinal disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal wall mass (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Buccal polyp (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Duodenal vascular ectasia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastric dysplasia (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrooesophagitis (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Ileal ulcer (Gastrointestinal disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 1 | 1
Internal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Lip haematoma (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1
Mouth cyst (Gastrointestinal disorders) | 0 | 1
Oedema mouth (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophageal dysplasia (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatic calcification (Gastrointestinal disorders) | 0 | 1
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Papilla of (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Spigelian hernia (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 64 | 67
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 33
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 21
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 21
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 17
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 10
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 9
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 10
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 9
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Metastases to lymph node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Non-Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hypopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Optic nerve neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Soft tissue cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testicular malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 55 | 46
Hypotension (Vascular disorders) | 39 | 27
Hypertension (Vascular disorders) | 32 | 29
Aortic aneurysm (Vascular disorders) | 24 | 35
Peripheral vascular disorder (Vascular disorders) | 27 | 24
Intermittent claudication (Vascular disorders) | 28 | 21
Peripheral artery stenosis (Vascular disorders) | 21 | 23
Peripheral ischaemia (Vascular disorders) | 20 | 19
Aortic stenosis (Vascular disorders) | 15 | 16
Hypertensive crisis (Vascular disorders) | 16 | 15
Haematoma (Vascular disorders) | 13 | 5
Femoral artery occlusion (Vascular disorders) | 12 | 5
Circulatory collapse (Vascular disorders) | 10 | 6
Orthostatic hypotension (Vascular disorders) | 8 | 7
Arteriosclerosis (Vascular disorders) | 6 | 7
Thrombosis (Vascular disorders) | 3 | 7
Hypovolaemic shock (Vascular disorders) | 2 | 6
Peripheral artery aneurysm (Vascular disorders) | 2 | 6
Peripheral artery thrombosis (Vascular disorders) | 5 | 3
Varicose vein (Vascular disorders) | 3 | 5
Iliac artery occlusion (Vascular disorders) | 7 | 0
Arterial stenosis (Vascular disorders) | 2 | 4
Aortic dissection (Vascular disorders) | 4 | 1
Extremity necrosis (Vascular disorders) | 1 | 4
Haemorrhage (Vascular disorders) | 3 | 2
Subclavian artery stenosis (Vascular disorders) | 4 | 1
Venous thrombosis (Vascular disorders) | 1 | 4
Aortic aneurysm rupture (Vascular disorders) | 1 | 3
Arterial occlusive disease (Vascular disorders) | 1 | 3
Diabetic vascular disorder (Vascular disorders) | 1 | 3
Thrombophlebitis (Vascular disorders) | 2 | 2
Ischaemia (Vascular disorders) | 2 | 1
Peripheral embolism (Vascular disorders) | 1 | 2
Shock (Vascular disorders) | 1 | 2
Shock haemorrhagic (Vascular disorders) | 1 | 2
Venous insufficiency (Vascular disorders) | 2 | 1
Accelerated hypertension (Vascular disorders) | 0 | 2
Aortic thrombosis (Vascular disorders) | 0 | 2
Arterial disorder (Vascular disorders) | 1 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 2 | 0
Subclavian artery occlusion (Vascular disorders) | 2 | 0
Venous stenosis (Vascular disorders) | 2 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0
Aneurysm ruptured (Vascular disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Aortic calcification (Vascular disorders) | 1 | 0
Aortic dilatation (Vascular disorders) | 1 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0
Arterial rupture (Vascular disorders) | 1 | 0
Artery dissection (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0
Extravasation blood (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Haematocoele (Vascular disorders) | 0 | 1
Hypoperfusion (Vascular disorders) | 0 | 1
Iliac artery rupture (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Ischaemic limb pain (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Renovascular hypertension (Vascular disorders) | 0 | 1
Subclavian artery aneurysm (Vascular disorders) | 1 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 1
Varicose ulceration (Vascular disorders) | 0 | 1
Varicose vein ruptured (Vascular disorders) | 0 | 1
Vascular insufficiency (Vascular disorders) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 28 | 19
Fall (Injury, poisoning and procedural complications) | 17 | 11
Femur fracture (Injury, poisoning and procedural complications) | 11 | 12
Hip fracture (Injury, poisoning and procedural complications) | 10 | 13
Subdural haematoma (Injury, poisoning and procedural complications) | 8 | 15
Femoral neck fracture (Injury, poisoning and procedural complications) | 12 | 6
Head injury (Injury, poisoning and procedural complications) | 11 | 7
Tendon rupture (Injury, poisoning and procedural complications) | 8 | 8
Rib fracture (Injury, poisoning and procedural complications) | 9 | 6
Laceration (Injury, poisoning and procedural complications) | 9 | 4
Ankle fracture (Injury, poisoning and procedural complications) | 7 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 5
Radius fracture (Injury, poisoning and procedural complications) | 5 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 5 | 5
Post procedural complication (Injury, poisoning and procedural complications) | 5 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 6
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 | 5
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 5
Toxicity to various agents (Injury, poisoning and procedural complications) | 6 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 8 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 6 | 3
Vascular graft occlusion (Injury, poisoning and procedural complications) | 8 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 5 | 3
Vascular graft complication (Injury, poisoning and procedural complications) | 6 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 | 3
Arterial restenosis (Injury, poisoning and procedural complications) | 4 | 3
Joint injury (Injury, poisoning and procedural complications) | 3 | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 4 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 5 | 2
Concussion (Injury, poisoning and procedural complications) | 4 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 4 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 4 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 4
Overdose (Injury, poisoning and procedural complications) | 5 | 1
Patella fracture (Injury, poisoning and procedural complications) | 4 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 4
Wound (Injury, poisoning and procedural complications) | 2 | 4
Alcohol poisoning (Injury, poisoning and procedural complications) | 4 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 2
Graft thrombosis (Injury, poisoning and procedural complications) | 2 | 2
Limb injury (Injury, poisoning and procedural complications) | 3 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 4 | 0
Injury (Injury, poisoning and procedural complications) | 3 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1
Thermal burn (Injury, poisoning and procedural complications) | 4 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 3 | 0
Arterial injury (Injury, poisoning and procedural complications) | 2 | 1
Burns second degree (Injury, poisoning and procedural complications) | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 3 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia, Obstruction (Injury, poisoning and procedural complications) | 3 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 2
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Bone contusion (Injury, poisoning and procedural complications) | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Liver contusion (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 2
Suture related complication (Injury, poisoning and procedural complications) | 1 | 1
Transplant failure (Injury, poisoning and procedural complications) | 2 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 2 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 2
Accident at home (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1
Internal injury (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Kidney contusion (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Testicular injury (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary bladder rupture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Venomous sting (Injury, poisoning and procedural complications) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 52 | 50
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 52
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 26 | 35
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 | 18
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20 | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 17
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 | 10
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 78 | 73
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 20
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 24 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 13
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 16 | 13
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 | 11
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 7
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 5
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 4 | 3
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 1
Articular calcification (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 61 | 83
Renal failure (Renal and urinary disorders) | 17 | 31
Haematuria (Renal and urinary disorders) | 15 | 12
Urinary retention (Renal and urinary disorders) | 19 | 7
Renal failure chronic (Renal and urinary disorders) | 13 | 10
Nephrolithiasis (Renal and urinary disorders) | 10 | 11
Renal impairment (Renal and urinary disorders) | 8 | 9
Calculus ureteric (Renal and urinary disorders) | 9 | 6
Renal colic (Renal and urinary disorders) | 8 | 6
Urethral stenosis (Renal and urinary disorders) | 5 | 5
Renal artery stenosis (Renal and urinary disorders) | 4 | 5
Hydronephrosis (Renal and urinary disorders) | 7 | 0
Acute prerenal failure (Renal and urinary disorders) | 3 | 3
Calculus urinary (Renal and urinary disorders) | 5 | 1
Renal cyst (Renal and urinary disorders) | 3 | 2
Renal tubular necrosis (Renal and urinary disorders) | 2 | 2
Calculus bladder (Renal and urinary disorders) | 2 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 2
Nephrotic syndrome (Renal and urinary disorders) | 0 | 3
Cystitis noninfective (Renal and urinary disorders) | 2 | 0
Micturition disorder (Renal and urinary disorders) | 2 | 0
Renal infarct (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 2
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 1
Bladder dysfunction (Renal and urinary disorders) | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 0 | 1
Cystitis glandularis (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Cystitis ulcerative (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis Chronic (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal artery dissection (Renal and urinary disorders) | 0 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 1 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0
Renal painr (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urethral disorder (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 37 | 27
Dehydration (Metabolism and nutrition disorders) | 24 | 33
Hypoglycaemia (Metabolism and nutrition disorders) | 26 | 24
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 | 26
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 10
Gout (Metabolism and nutrition disorders) | 5 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 4 | 2
Obesity (Metabolism and nutrition disorders) | 2 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Fructose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 28 | 30
Cholecystitis acute (Hepatobiliary disorders) | 24 | 19
Cholecystitis chronic (Hepatobiliary disorders) | 7 | 5
Bile duct stone (Hepatobiliary disorders) | 3 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 5
Cholangitis (Hepatobiliary disorders) | 3 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 3
Biliary colic (Hepatobiliary disorders) | 1 | 3
Hepatic steatosis (Hepatobiliary disorders) | 3 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 3
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 2 | 0
Cholestasish (Hepatobiliary disorders) | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 2
Hepatitis alcoholic (Hepatobiliary disorders) | 2 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Portal hypertension (Hepatobiliary disorders) | 2 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary fistula (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 3
Pneumobilia (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 52 | 42
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 5
Coagulopathy (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Bone marrow ischaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hyperprothrombinaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Jaundice acholuric (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 28 | 31
Prostatitis (Reproductive system and breast disorders) | 4 | 9
Prostatomegaly (Reproductive system and breast disorders) | 8 | 2
Ovarian cyst (Reproductive system and breast disorders) | 2 | 3
Uterine polyp (Reproductive system and breast disorders) | 2 | 3
Acquired phimosis (Reproductive system and breast disorders) | 2 | 2
Uterine prolapse (Reproductive system and breast disorders) | 2 | 2
Epididymitis (Reproductive system and breast disorders) | 1 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 1
Epididymal cyst (Reproductive system and breast disorders) | 2 | 0
Scrotal oedema (Reproductive system and breast disorders) | 2 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Genital pain (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1
Peyronie's disease (Reproductive system and breast disorders) | 1 | 0
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal polyp (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 11 | 4
Hepatic enzyme increased (Investigations) | 5 | 8
International normalised ratio increased (Investigations) | 5 | 3
Weight decreased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 1
Liver function test abnormal (Investigations) | 2 | 5
Blood bilirubin increased (Investigations) | 2 | 4
Troponin increased (Investigations) | 3 | 3
Blood creatinine increased (Investigations) | 4 | 1
Blood glucose increased (Investigations) | 3 | 2
Haemoglobin decreased (Investigations) | 1 | 4
Blood pressure increased (Investigations) | 1 | 3
Ejection fraction decreased (Investigations) | 4 | 0
Electrocardiogram ST segment depression (Investigations) | 3 | 0
Prostatic specific antigen increased (Investigations) | 1 | 2
Blood potassium decreased (Investigations) | 2 | 0
Blood pressure decreased (Investigations) | 0 | 2
Cardiac stress test abnormal (Investigations) | 0 | 2
Heart rate decreased (Investigations) | 1 | 1
Heart rate irregular (Investigations) | 2 | 0
Intraocular pressure increased (Investigations) | 1 | 1
Troponin I increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 1
Aspartate aminotransferase abnormal (Investigations) | 0 | 1
Bile output abnormal (Investigations) | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Carotid bruit (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 0 | 1
Streptococcus test positive (Investigations) | 0 | 1
Stroke volume decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 12 | 8
Depression (Psychiatric disorders) | 7 | 8
Delirium (Psychiatric disorders) | 4 | 7
Mental status changes (Psychiatric disorders) | 6 | 2
Anxiety (Psychiatric disorders) | 4 | 2
Suicide attempt (Psychiatric disorders) | 1 | 5
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 | 3
Completed suicide (Psychiatric disorders) | 3 | 2
Alcohol abuse (Psychiatric disorders) | 2 | 2
Anxiety disorder (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Major depression (Psychiatric disorders) | 2 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 1
Conversion disorder (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 1
Suicidal behaviour (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Dysthymic disorder (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Impulse-control disorder (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Psychogenic seizure (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 | 1
Cataract (Eye disorders) | 16 | 16
Retinal detachment (Eye disorders) | 3 | 3
Amaurosis fugax (Eye disorders) | 3 | 1
Vitreous haemorrhage (Eye disorders) | 2 | 2
Diabetic retinopathy (Eye disorders) | 0 | 3
Diplopia (Eye disorders) | 1 | 2
Glaucoma (Eye disorders) | 1 | 2
Blindness (Eye disorders) | 1 | 1
Ocular vascular disorder (Eye disorders) | 1 | 1
Retinal artery occlusion (Eye disorders) | 0 | 2
Retinal ischaemia (Eye disorders) | 0 | 2
Retinal tear (Eye disorders) | 2 | 0
Retinal vein occlusion (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1
Diabetic eye disease (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Ocular retrobulbar haemorrhag (Eye disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 14 | 5
Ophthalmoplegia (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 8 | 5
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 14
Vestibular disorder (Ear and labyrinth disorders) | 4 | 2
Vertigo positional (Ear and labyrinth disorders) | 3 | 1
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 1
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Ototoxicity (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 4 | 4
Goitre (Endocrine disorders) | 2 | 3
Adrenal disorder (Endocrine disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 5 | 6
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 2
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 | 1
Spinal vessel congenital anomaly (Congenital, familial and genetic disorders) | 0 | 1
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 4
Allergy to arthropod sting (Immune system disorders) | 3 | 1
Hypersensitivity (Immune system disorders) | 2 | 2
Allergy to arthropod bite (Immune system disorders) | 1 | 1
Allergic oedema (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Disability (Social circumstances) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 1 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 17 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7890) | Darapladib (N=7912)
Anaemia (Blood and lymphatic system disorders) | 208 | 191
Angina pectoris (Cardiac disorders) | 528 | 457
Atrial fibrillation (Cardiac disorders) | 245 | 257
Cataract (Eye disorders) | 198 | 203
Abdominal pain (Gastrointestinal disorders) | 188 | 163
Abdominal pain upper (Gastrointestinal disorders) | 152 | 180
Abnormal faeces (Gastrointestinal disorders) | 63 | 728
Constipation (Gastrointestinal disorders) | 255 | 247
Diarrhoea (Gastrointestinal disorders) | 479 | 949
Dyspepsia (Gastrointestinal disorders) | 182 | 177
Flatulence (Gastrointestinal disorders) | 92 | 189
Gastritis (Gastrointestinal disorders) | 192 | 159
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 160 | 144
Large intestine polyp (Gastrointestinal disorders) | 265 | 259
Nausea (Gastrointestinal disorders) | 222 | 228
Fatigue (General disorders) | 357 | 354
Non-cardiac chest pain (General disorders) | 376 | 366
Oedema peripheral (General disorders) | 419 | 431
Bronchitis (Infections and infestations) | 416 | 389
Influenza (Infections and infestations) | 253 | 223
Nasopharyngitis (Infections and infestations) | 588 | 548
Sinusitis (Infections and infestations) | 189 | 157
Upper respiratory tract infection (Infections and infestations) | 425 | 367
Urinary tract infection (Infections and infestations) | 296 | 260
Blood glucose increased (Investigations) | 181 | 171
Blood pressure increased (Investigations) | 197 | 173
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 608 | 566
Arthralgia (Musculoskeletal and connective tissue disorders) | 401 | 385
Back pain (Musculoskeletal and connective tissue disorders) | 466 | 421
Muscle spasms (Musculoskeletal and connective tissue disorders) | 168 | 164
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 219 | 180
Myalgia (Musculoskeletal and connective tissue disorders) | 244 | 207
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 176 | 167
Pain in extremity (Musculoskeletal and connective tissue disorders) | 354 | 315
Dizziness (Nervous system disorders) | 491 | 456
Headache (Nervous system disorders) | 357 | 296
Insomnia (Psychiatric disorders) | 164 | 126
Urine odour abnormal (Renal and urinary disorders) | 81 | 473
Cough (Respiratory, thoracic and mediastinal disorders) | 404 | 401
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 346 | 324
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 34 | 383
Hypertension (Vascular disorders) | 660 | 643
Hypotension (Vascular disorders) | 181 | 184

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.